CLINICAL TRIAL: NCT00262028
Title: A Phase 2, Randomized, Single-blind, Controlled, Single-Center Study to Compare the Safety and Immunogenicity of One Dose of Chiron Meningococcal ACWY Conjugate Vaccine With One Dose of Licensed Meningococcal ACWY Polysaccharide Vaccine Administered to Healthy Children 2-10 Years of Age and an Open-label Study to Assess the Safety and Immunogenicity of One Dose of Chiron Meningococcal ACWY Conjugate Vaccine Administered to Healthy Toddlers 12-23 Months of Age
Brief Title: Study of the Safety and Immune Response of a Meningococcal Vaccine Administered to Healthy Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V59P8
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Prevention of Meningococcal Disease
MeSH Terms: interventions — MenACWY-CRM vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- MenACWY-CRM (2-10 years) (Experimental): Subjects received one dose of investigational MenACWY-CRM conjugate vaccine
  Interventions: Biological: MenACWY-CRM Vaccine
- MenACWY-CRM (12-23 months) (Experimental): Subjects received one dose of investigational MenACWY-CRM conjugate vaccine
  Interventions: Biological: MenACWY-CRM Vaccine
- MenACWY-PS (2-10 years) (Active Comparator): Subjects received one dose of licensed comparator MenACWY polysaccharide (MenACWY-PS) vaccine
  Interventions: Biological: MenACWY-PS Vaccine
- MenACWY-CRM+PnC (12-15 months) (Experimental): Subjects received one dose of MenACWY-CRM vaccine alone or concomitantly with PnC
  Interventions: Biological: MenACWY-CRM Vaccine
- MenACWY-CRM+DTaP (16-23 months) (Experimental): Subjects received one dose of MenACWY-CRM vaccine alone or concomitantly with DTaP
  Interventions: Biological: MenACWY-CRM Vaccine

INTERVENTIONS:
Biological: MenACWY-CRM Vaccine
  Arms: MenACWY-CRM (12-23 months); MenACWY-CRM (2-10 years); MenACWY-CRM+DTaP (16-23 months); MenACWY-CRM+PnC (12-15 months)
Biological: MenACWY-PS Vaccine
  Arms: MenACWY-PS (2-10 years)

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of Novartis (formerly Chiron) Meningococcal ACWY Conjugate Vaccine administered to healthy children ages 1 - 10 years

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Healthy children 2-10 years of age;
* Group 2: Healthy toddlers 12-23 months of age; who are up to date with age appropriate immunizations for diphtheria, tetanus, pertussis, polio, hepatitis B, Hemophilus influenzae type b, and pneumococcus.

Exclusion Criteria:

* Group 1: Subjects with a previous or suspected disease caused by N. meningitidis; or previous immunization with a meningococcal vaccine or vaccine containing meningococcal antigen(s); Any serious acute, chronic or progressive disease.
* Group 2: Subjects with a previous or suspected disease caused by N. meningitidis or previous immunization with a meningococcal vaccine or vaccine containing meningococcal antigen(s); Any serious acute, chronic or progressive disease.

Ages: 12 Months to 10 Years | Sex: All
Age Groups: Child
Enrollment: 910 (Actual)
Dates: Start 2005-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines & Diagnostics
Locations (1):
- Kaiser Permanente Vaccine Study Center, Oakland, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a single center.
Pre-assignment Details: All enrolled subjects participated in this study.
Groups:
- MenACWY (2-5 Years Old): Subjects received one dose of the investigational MenACWY-cross-reactive material (CRM) conjugate vaccine.
- MenACWY-PS (2-5 Years Old); MenACWY-PS (6-10 Years Old): Subjects received one dose of the licensed MenACWY-polysaccharide vaccine.
- MenACWY (6-10 Years Old); MenACWY (12-15 Months Old); MenACWY (16-23 Months): Subjects received one dose of the investigational MenACWY-CRM conjugate vaccine.
- MenACWY+PnC (12-15 Months): Subjects received one dose of the MenACWY-CRM conjugate vaccine administered concomitantly with pneumococcal conjugate vaccine (PnC).
- MenACWY+DTaP (16-23 Months): Subjects received one dose of the MenACWY-CRM conjugate vaccine administered concomitantly with diphtheria-tetanus-acellular pertussis (DTaP) vaccine.
- MenACWY-PS (3-5 Years Old): Children aged 3 to 5 years receiving MenACWY- polysaccharide (PS) vaccine from the first part of the study (Menomune, not licensed in US in children under 2 years of age) were used as controls for the 12-23-months-old part two toddlers.
Period: Overall Study
Arm/Group | MenACWY (2-5 Years Old) | MenACWY-PS (2-5 Years Old) | MenACWY (6-10 Years Old) | MenACWY-PS (6-10 Years Old) | MenACWY (12-15 Months Old) | MenACWY+PnC (12-15 Months) | MenACWY (16-23 Months) | MenACWY+DTaP (16-23 Months) | MenACWY-PS (3-5 Years Old)
Started | 152 | 153 | 157 | 157 | 74 | 73 | 71 | 73 | 100
Completed | 128 | 126 | 137 | 134 | 62 | 60 | 59 | 55 | 81
Not Completed | 24 | 27 | 20 | 23 | 12 | 13 | 12 | 18 | 19
Not completed — Withdrawal by Subject | 6 | 3 | 6 | 5 | 2 | 3 | 5 | 7 | 2
Not completed — Lost to Follow-up | 7 | 7 | 5 | 5 | 4 | 3 | 3 | 5 | 6
Not completed — Administrative Reason | 11 | 14 | 9 | 12 | 6 | 7 | 4 | 6 | 10
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Unable to classify | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- MenACWY (2-5 Years Old); MenACWY (6-10 Years Old); MenACWY (12-15 Months Old); MenACWY (16-23 Months Old): Subjects received one dose of the investigational MenACWY-CRM conjugate vaccine.
- MenACWY-PnC (12-15 Months Old): Subjects received one dose of the MenACWY-CRM conjugate vaccine administered concomitantly with pneumococcal conjugate vaccine.
- MenACWY+DTaP (16-23 Months Old): Subjects received one dose of the MenACWY-CRM conjugate vaccine administered concomitantly with DTaP vaccine.
- MenACWY+PS (3-5 YearsOld): Children aged 3 to 5 years receiving MenACWY-PS from the first part of the study (Menomune, not licensed in US in children under 2 years of age) were used as controls for the 12-23-months-old part two toddlers.
- Total: Total of all reporting groups
Arm/Group | MenACWY (2-5 Years Old) | MenACWY-PS (2-5 Years Old) | MenACWY (6-10 Years Old) | MenACWY-PS (6-10 Years Old) | MenACWY (12-15 Months Old) | MenACWY-PnC (12-15 Months Old) | MenACWY (16-23 Months Old) | MenACWY+DTaP (16-23 Months Old) | MenACWY+PS (3-5 YearsOld) | Total
Number analyzed (Participants) | 152 | 153 | 157 | 157 | 74 | 73 | 71 | 73 | 100 | 1010
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.3 (1.2) | 3.3 (1.2) | 8.0 (1.5) | 8.0 (1.4) | NA (NA) — Data are reported in a separate table | NA (NA) — Data are reported in a separate table | NA (NA) — Data are reported in a separate table | NA (NA) — Data are reported in a separate table | NA (NA) — Data are reported in a separate table | 5.7 (2.7)
Age, Continuous [Mean (Standard Deviation); unit: months] | NA (NA) — Data are reported in the previous table | NA (NA) — Data are reported in the previous table | NA (NA) — Data are reported in the previous table | NA (NA) — Data are reported in the previous table | 12.2 (0.5) | 12.2 (0.5) | 18.2 (1.3) | 18.2 (1.4) | 52.6 (11.4) | 24.7 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 79 | 80 | 78 | NA — Data are reported in a separate table | NA — reported in a separate table | NA — reported in a separate table | NA — reported in a separate table | NA — reported in a separate table | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 86 | 74 | 77 | 79 | NA — reported in a separate table | NA — reported in a separate table | NA — reported in a separate table | NA — reported in a separate table | NA — reported in a separate table | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data are reported in the previous table | NA — Data are reported in the previous table | NA — Data are reported in the previous table | NA — Data are reported in the previous table | 30 | 29 | 31 | 36 | 51 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data are reported in the previous table | NA — Data are reported in the previous table | NA — Data are reported in the previous table | NA — Data are reported in the previous table | 44 | 44 | 40 | 37 | 49 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects (2-10 Years of Age) With Human Serum Bactericidal Activity (hSBA) Titers ≥1:4 After Receiving Either MenACWY-CRM or MenACWY-PS Vaccine
Description: Number of subjects (2-10 years of age) achieving with hSBA titers ≥1:4 against Neisseria meningitidis serogroups A,C,W and Y, one month after receiving one dose of either MenACWY-CRM vaccine or MenACWY-PS vaccine.
Time Frame: 1 month post vaccination (Day 29)
Population: Analysis was done on per protocol population i.e. all subjects who received one dose of vaccine and provided serum samples at the relevant time points (day 1, day 29 and day 360) and had no major protocol deviation.
Measure: Number; unit: Subjects
Groups:
- MenACWY-CRM (2-10 Years Old): Subjects received one dose of the investigational MenACWY-CRM conjugate vaccine
- MenACWY-PS (2-10 Years): Subjects received one dose of the licensed MenACWY-PS vaccine
Arm/Group | MenACWY-CRM (2-10 Years Old) | MenACWY-PS (2-10 Years)
Number analyzed (Participants) | 284 | 285
Subjects
  Serogroup A (Day 1), N=280, 281 | 6 | 1
  Serogroup A (Day 29), N=280, 281 | 228 | 125
  Serogroup C (Day 1) | 80 | 81
  Serogroup C (Day 29) | 232 | 181
  Serogroup W (Day 1), N=279, 282 | 111 | 108
  Serogroup W (Day 29), N=279, 282 | 263 | 202
  Serogroup Y (Day 1), N=280, 282 | 61 | 68
  Serogroup Y (Day 29), N=280, 282 | 254 | 167
Statistical Analysis 1: Comparison: MenACWY-CRM (2-10 Years Old) vs MenACWY-PS (2-10 Years); Noninferiority of immune responses of MenACWY-CRM to licensed comparator against serogroup A; Test type: Non-Inferiority or Equivalence — MenACWY-CRM was considered to be noninferior to the licensed comparator if the lower limit (LL) of the 95% confidence intervals (CI) of the difference (MenACWY minus licensed comparator)in the percentage of the subjects with hSBA titer ≥ 1:4 at one month post vaccination was > -10% against each serogroup; Vaccine group difference = 37, 95% CI 2-sided [29 to 44]
Statistical Analysis 2: Comparison: MenACWY-CRM (2-10 Years Old) vs MenACWY-PS (2-10 Years); Noninferiority of immune responses of MenACWY-CRM to licensed comparator against serogroup C; Test type: Non-Inferiority or Equivalence — MenACWY-CRM was considered to be noninferior to the licensed comparator if the lower LL of the 95% CI of the difference (MenACWY minus licensed comparator)in the percentage of the subjects with hSBA titer ≥ 1:4 at one month post vaccination was > -10% against each serogroup; Vaccine group difference = 19, 95% CI 2-sided [12 to 26]
Statistical Analysis 3: Comparison: MenACWY-CRM (2-10 Years Old) vs MenACWY-PS (2-10 Years); Noninferiority of immune responses of MenACWY-CRM to licensed comparator against serogroup W; Test type: Non-Inferiority or Equivalence — MenACWY-CRM was considered to be noninferior to the licensed comparator if the LL of the 95% CI of the difference (MenACWY minus licensed comparator)in the percentage of the subjects with hSBA titer ≥ 1:4 at one month post vaccination was > -10% against each serogroup; Vaccine group difference = 23, 95% CI 2-sided [17 to 29]
Statistical Analysis 4: Comparison: MenACWY-CRM (2-10 Years Old) vs MenACWY-PS (2-10 Years); No inferiority of immune responses of MenACWY-CRM to licensed comparator against serogroup Y; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; Vaccine group difference = 31, 95% CI 2-sided [25 to 38]
Statistical Analysis 5: Comparison: MenACWY-CRM (2-10 Years Old) vs MenACWY-PS (2-10 Years); Superiority of immune responses of MenACWY-CRM to licensed comparator against serogroup A MenACWY-CRM was considered to be superior to the licensed comparator if the LL of the 95% CI of the difference (MenACWY minus licensed comparator) in the percentage of the subjects with hSBA titer ≥ 1:4 at one month post vaccination was > 0% against each serogroup; Test type: Superiority or Other; Vaccine group difference = 37, 95% CI 2-sided [29 to 44]
Statistical Analysis 6: Comparison: MenACWY-CRM (2-10 Years Old) vs MenACWY-PS (2-10 Years); Superiority of immune responses of MenACWY-CRM to licensed comparator against serogroup C MenACWY-CRM was considered to be superior to the licensed comparator if the LL of the 95% CI of the difference (MenACWY minus licensed comparator) in the percentage of the subjects with hSBA titer ≥ 1:4 at one month post vaccination was > 0% against each serogroup; Test type: Superiority or Other; Vaccine group difference = 19, 95% CI 2-sided [12 to 26]
Statistical Analysis 7: Comparison: MenACWY-CRM (2-10 Years Old) vs MenACWY-PS (2-10 Years); Superiority of immune responses of MenACWY-CRM to licensed comparator against serogroup W MenACWY-CRM was considered to be superior to the licensed comparator if the LL of the 95% CI of the difference (MenACWY minus licensed comparator) in the percentage of the subjects with hSBA titer ≥ 1:4 at one month post vaccination was > 0% against each serogroup; Test type: Superiority or Other; Vaccine group difference = 23, 95% CI 2-sided [17 to 29]
Statistical Analysis 8: Comparison: MenACWY-CRM (2-10 Years Old) vs MenACWY-PS (2-10 Years); Superiority of immune responses of MenACWY-CRM to licensed comparator against serogroup Y MenACWY-CRM was considered to be superior to the licensed comparator if the LL of the 95% CI of the difference (MenACWY minus licensed comparator) in the percentage of the subjects with hSBA titer ≥ 1:4 at one month post vaccination was > 0% against each serogroup; Test type: Superiority or Other; Vaccine group difference = 31, 95% CI 2-sided [25 to 38]

2. Secondary Outcome: Percentages of Subjects (2-5 Years of Age and 6-10 Years of Age) With hSBA ≥ 1:4 After Receiving Either MenACWY-CRM or MenACWY-PS Vaccine
Description: Percentages of subjects (2-5 years of age and 6-10 years of age) with hSBA ≥ 1:4 directed against N. meningitidis serogroups A, C, W and Y, one month after receiving one dose of either MenACWY-CRM vaccine or MenACWY-PS vaccine.
Time Frame: 1 month post vaccination (Day 29)
Population: Analysis was done on per protocol population. The total number of participants analyzed in the MenACWY-CRM (2-10 Years Old) group (282), is different respect with that reported in the Outcome Measure 1 (281). There, the largest number for each group across the 4 strains was reported (not all strains had a result from the lab-i.e. C strain).
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- MenACWY-CRM (2-5 Years Old): Subjects received one dose of the investigational MenACWY-CRM conjugate vaccine
- MenACWY-PS (2-5 Years Old): Subjects received one dose of the licensed MenACWY-PS vaccine
- MenACWY-CRM (6-10 Years Old): Subjects received one dose of investigational MenACWY-CRM vaccine
- MenACWY-PS (6-10 Years Old): Subjects received one dose of licensed MenACWY-PS vaccine
Arm/Group | MenACWY-CRM (2-5 Years Old) | MenACWY-PS (2-5 Years Old) | MenACWY-CRM (6-10 Years Old) | MenACWY-PS (6-10 Years Old)
Number analyzed (Participants) | 135 | 138 | 147 | 145
Percentages of subjects
  Serogroup A (Day 1), N=133,138,147,143 | 2 [0 to 5] | 0 [0 to 3] | 3 [1 to 7] | 1 [0.018 to 4]
  Serogroup A (Day 29), N=133,138,147,143 | 80 [72 to 86] | 43 [34 to 51] | 83 [76 to 89] | 46 [38 to 55]
  Serogroup C (Day 1), N=135,138,146,145 | 23 [16 to 31] | 11 [6 to 17] | 34 [26 to 42] | 46 [37 to 54]
  Serogroup C (Day 29), N=135,138,146,145 | 76 [68 to 83] | 45 [36 to 54] | 88 [82 to 93] | 82 [75 to 88]
  Serogroup W (Day 1), N=135,138,144,144 | 32 [24 to 40] | 22 [16 to 30] | 47 [39 to 56] | 53 [45 to 62]
  Serogroup W (Day 29), N=135,138,144,144 | 90 [84 to 95] | 55 [46 to 64] | 98 [94 to 100] | 88 [81 to 92]
  Serogroup Y (Day 1), N=134,138,146,144 | 18 [12 to 25] | 13 [8 to 20] | 25 [19 to 33] | 35 [27 to 43]
  Serogroup Y (Day 29), N=134,138,146,144 | 87 [80 to 92] | 49 [40 to 57] | 95 [89 to 98] | 69 [61 to 77]

3. Secondary Outcome: Percentages of Subjects (12-23 Months Old) With hSBA Titer ≥ 1:4 After Receiving MenACWY-CRM Vaccine Compared With Percentage of Subjects (3-5 Years Old) With hSBA Titer ≥ 1:4 After Receiving MenACWY-PS Vaccine
Description: Percentage of subjects (12-23 months old) with hSBA ≥ 1:4 directed against N. meningitidis serogroups A, C, W and Y after receiving one dose of MenACWY-CRM vaccine compared with percentage of subjects (3-5 years old) with hSBA ≥ 1:4 after one dose of licensed MenACWY-PS vaccine.
Time Frame: 1 month post vaccination (Day 29)
Population: Analysis was done on per protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- MenACWY-CRM (12-23 Months Old): Subjects received one dose of the investigational MenACWY-CRM conjugate vaccine
- MenACWY-PS (3-5 Years Old): Subjects received one dose of the licensed MenACWY-PS vaccine. This group was a subset of the licensed comparator (2-5 years old) cohort that received one dose of licensed MenACWY-PS vaccine
Arm/Group | MenACWY-CRM (12-23 Months Old) | MenACWY-PS (3-5 Years Old)
Number analyzed (Participants) | 241 | 91
Percentages of subjects
  Serogroup A (Day 1), N=240,91 | 0 [0 to 2] | 0 [0 to 4]
  Serogroup A (Day 29), N=240,91 | 81 [76 to 86] | 51 [40 to 61]
  Serogroup C (Day 1), N=241,91 | 3 [1 to 6] | 12 [6 to 21]
  Serogroup C (Day 29), N=241,91 | 90 [86 to 94] | 42 [32 to 53]
  Serogroup W (Day 1), N=240,91 | 3 [1 to 6] | 24 [16 to 34]
  Serogroup W (Day 29), N=240,91 | 86 [81 to 90] | 63 [52 to 73]
  Serogroup Y (Day 1), N=238,91 | 2 [1 to 5] | 15 [9 to 24]
  Serogroup Y (Day 29), N=238,91 | 64 [58 to 70] | 51 [40 to 61]

4. Secondary Outcome: hSBA Geometric Mean Titer (GMT) in Subjects (2-10 Years of Age) After Receiving Either MenACWY-CRM Vaccine or MenACWY-PS Vaccine
Description: hSBA GMT against N. meningitidis serogroups A, C, W, and Y, in subjects (2-10 years of age), one month after receiving one dose of either MenACWY-CRM vaccine or the licensed MenACWY-PS vaccine.
Time Frame: 1 month post vaccination (Day 29)
Population: Analysis was done on per protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM (2-10 Years Old) | MenACWY-PS (2-10 Years)
Number analyzed (Participants) | 281 | 283
Titers
  Serogroup A (Day 1), N=280, 281 | 2.06 [2.02 to 2.1] | 2.02 [1.98 to 2.06]
  Serogroup A (Day 29), N=280, 281 | 36 [30 to 44] | 6.31 [5.21 to 7.64]
  Serogroup C (Day 1) | 3.07 [2.77 to 3.4] | 3.33 [3.01 to 3.68]
  Serogroup C (Day 29) | 26 [21 to 34] | 15 [12 to 20]
  Serogroup W (Day 1), N=279, 282 | 5.74 [4.86 to 6.78] | 5.63 [4.77 to 6.65]
  Serogroup W (Day 29), N=279, 282 | 60 [50 to 71] | 14 [12 to 17]
  Serogroup Y (Day 1), N=280, 282 | 3.32 [2.95 to 3.73] | 3.34 [2.97 to 3.76]
  Serogroup Y (Day 29), N=280, 282 | 54 [44 to 66] | 11 [9.29 to 14]

5. Secondary Outcome: hSBA GMT in Subjects (2-5 Years of Age and 6-10 Years of Age) Receiving Either MenACWY-CRM Vaccine or MenACWY-PS Vaccine
Description: hSBA GMT against N. meningitidis serogroups A, C, W, and Y, in subjects (2-5 years of age and 6-10 years of age), one month after receiving one dose of either MenACWY-CRM vaccine or licensed MenACWY-PS vaccine.
Time Frame: 1 month post vaccination (Day 29)
Population: Analysis was done on per protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- MenACWY-PS (2-5 Years Old): Subjects received one dose of the MenACWY-PS vaccine
- MenACWY-CRM (6-10 Years Old): Subjects received one dose of MenACWY-CRM conjugate vaccine
- MenACWY-PS (6-10 Years Old): Subjects received one dose of MenACWY-PS vaccine
Arm/Group | MenACWY-CRM (2-5 Years Old) | MenACWY-PS (2-5 Years Old) | MenACWY-CRM (6-10 Years Old) | MenACWY-PS (6-10 Years Old)
Number analyzed (Participants) | 135 | 138 | 147 | 145
Titer
  Serogroup A (Day 1), N=133,138,147,143 | 2.04 [2 to 2.07] | 2 [1.97 to 2.03] | 2.08 [2.01 to 2.15] | 2.03 [1.96 to 2.11]
  Serogroup A (Day 29), N=133,138,147,143 | 28 [22 to 37] | 5.8 [4.49 to 7.5] | 45 [34 to 60] | 6.84 [5.17 to 9.06]
  Serogroup C (Day 1), N=135,138,146,145 | 2.81 [2.52 to 3.13] | 2.38 [2.14 to 2.65] | 3.33 [2.84 to 3.9] | 4.58 [3.91 to 5.38]
  Serogroup C (Day 29), N=135,138,146,145 | 14 [11 to 19] | 6.93 [5.22 to 9.18] | 47 [34 to 67] | 33 [23 to 47]
  Serogroup W (Day 1), N=135,138,144,144 | 4.68 [3.78 to 5.8] | 3.64 [2.95 to 4.5] | 6.94 [5.45 to 8.84] | 8.55 [6.71 to 11]
  Serogroup W (Day 29), N=135,138,144,144 | 43 [34 to 56] | 7.84 [6.12 to 10] | 80 [65 to 99] | 24 [20 to 30]
  Serogroup Y (Day 1), N=134,138,146,144 | 3 [2.61 to 3.44] | 2.57 [2.24 to 2.95] | 3.65 [3.03 to 4.38] | 4.3 [3.58 to 5.18]
  Serogroup Y (Day 29), N=134,138,146,144 | 42 [31 to 56] | 7.17 [5.37 to 9.58] | 68 [51 to 90] | 18 [13 to 24]

6. Secondary Outcome: hSBA Geometric Mean Titer (GMT) in Subjects (12-23 Months Old) After Receiving MenACWY-CRM Vaccine Compared With hSBA GMT in 3-5 Year Old Subjects After Receiving MenACWY-PS Vaccine
Description: hSBA GMT against N. meningitidis serogroups A, C, W, and Y, in subjects (12-23 months old), one month after receiving one dose of MenACWY-CRM vaccine compared with hSBA GMT in 3-5 year old subjects after receiving one dose of licensed MenACWY-PS vaccine.
Time Frame: 1 month post vaccination (Day 29)
Population: Analysis was done on per protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- MenACWY-PS (3-5 Years Old): Subjects received one dose of the licensed MenACWY-PS vaccine This group was a subset of the Licensed comparator (2-5 year old) cohort that received one dose of licensed MenACWY-PS vaccine.
Arm/Group | MenACWY-CRM (12-23 Months Old) | MenACWY-PS (3-5 Years Old)
Number analyzed (Participants) | 241 | 91
Titer
  Serogroup A (Day 1), N=240,91 | 2 [2 to 2] | 2 [2 to 2]
  Serogroup A (Day 29), N=240,91 | 18 [15 to 21] | 7.18 [5.34 to 9.64]
  Serogroup C (Day 1), N=241,91 | 2.13 [2.02 to 2.25] | 2.44 [2.23 to 2.68]
  Serogroup C (Day 29), N=241,91 | 22 [18 to 26] | 7.09 [5.29 to 9.5]
  Serogroup W (Day 1), N=240,91 | 2.13 [1.94 to 2.33] | 3.91 [3.36 to 4.55]
  Serogroup W (Day 29), N=240,91 | 18 [15 to 21] | 9.52 [7.21 to 13]
  Serogroup Y (Day 1), N=238,91 | 2.11 [1.97 to 2.25] | 2.69 [2.42 to 3]
  Serogroup Y (Day 29), N=238,91 | 11 [8.91 to 14] | 8.48 [6.01 to 12]

7. Secondary Outcome: Number of Subjects (2-10 Years, 2-5 Years and 6-10 Years Old) With hSBA ≥ 1:4 After Receiving Either MenACWY-CRM Vaccine or MenACWY-PS Vaccine
Description: Number of subjects (2-10 years, 2-5 years and 6-10 years old subjects) with hSBA ≥ 1:4 directed against N. meningitidis serogroups A, C, W and Y, 12 months after receiving one dose of either MenACWY-CRM vaccine or MenACWY-PS vaccine.
Time Frame: 12 months post vaccination (Day 360)
Population: Analysis was done on per protocol population.
Measure: Number; unit: Subjects
Groups:
- MenACWY-CRM (2-5 Years); MenACWY-CRM (6-10 Years): Subjects received one dose of the investigational MenACWY-CRM conjugate vaccine
- MenACWY-PS (2-5 Years); MenACWY-PS (6-10 Years): Subjects received one dose of the licensed MenACWY-PS vaccine
Arm/Group | MenACWY-CRM (2-10 Years Old) | MenACWY-PS (2-10 Years) | MenACWY-CRM (2-5 Years) | MenACWY-PS (2-5 Years) | MenACWY-CRM (6-10 Years) | MenACWY-PS (6-10 Years)
Number analyzed (Participants) | 253 | 240 | 119 | 114 | 134 | 126
Subjects
  Serogroup A (Day 1), N=253,238,119,114,134,124 | 6 | 1 | 2 | 0 | 4 | 1
  Serogroup A (Day 360), N=253,238,119,114,134,124 | 71 | 44 | 27 | 15 | 44 | 29
  Serogroup C (Day 1), N=252,240,119,114,133,126 | 70 | 72 | 26 | 12 | 44 | 60
  Serogroup C (Day 360), N=252,240,119,114,133,126 | 172 | 126 | 77 | 41 | 95 | 85
  Serogroup W (Day 1), N=249,237,119,113,130,124 | 96 | 85 | 35 | 21 | 61 | 64
  Serogroup W (Day 360), N=249,237,119,113,130,124 | 234 | 119 | 108 | 41 | 126 | 78
  Serogroup Y (Day 1), N=250,239,118,113,132,126 | 53 | 59 | 22 | 14 | 31 | 45
  Serogroup Y (Day 360), N=250,239,118,113,132,126 | 215 | 90 | 101 | 26 | 114 | 64

8. Secondary Outcome: hSBA Geometric Mean Titer (GMT) in Subjects (2-10 Years, 2-5 Years and 6-10 Years Old) After Receiving Either MenACWY-CRM Vaccine or MenACWY-PS Vaccine
Description: hSBA GMT against N. meningitidis serogroups A, C, W, and Y, in subjects (2-10 years, 2-5 years and 6-10 years old), twelve months after receiving one dose of either MenACWY-CRM vaccine or MenACWY-PS vaccine.
Time Frame: 12 months post vaccination (Day 360)
Population: Analysis was done on per protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- MenACWY-PS (2-10 Years Old); MenACWY-PS (2-5 Years Old); MenACWY-PS (6-10 Years Old): Subjects received one dose of the licensed MenACWY-PS vaccine
- MenACWY-CRM (6-10 Years Old): Subjects received one dose of the investigational MenACWY-CRM conjugate vaccine
Arm/Group | MenACWY-CRM (2-10 Years Old) | MenACWY-PS (2-10 Years Old) | MenACWY-CRM (2-5 Years Old) | MenACWY-PS (2-5 Years Old) | MenACWY-CRM (6-10 Years Old) | MenACWY-PS (6-10 Years Old)
Number analyzed (Participants) | 253 | 240 | 119 | 114 | 134 | 126
Titer
  Serogroup A (Day 1), N=253,238,119,114,134,124 | 2.06 [2.02 to 2.11] | 2.02 [1.97 to 2.07] | 2.04 [2 to 2.08] | 2 [1.96 to 2.04] | 2.09 [2 to 2.17] | 2.04 [1.95 to 2.12]
  Serogroup A (Day 360), N=253,238,119114,134,124 | 3.88 [3.39 to 4.44] | 3 [2.61 to 3.44] | 3.15 [2.73 to 3.64] | 2.49 [2.15 to 2.89] | 4.66 [3.75 to 5.8] | 3.55 [2.83 to 4.45]
  Serogroup C (Day 1), N=252,240,119,114,133,126 | 3.04 [2.73 to 3.39] | 3.43 [3.07 to 3.84] | 2.77 [2.47 to 3.12] | 2.38 [2.11 to 2.69] | 3.3 [2.79 to 3.9] | 4.77 [4.01 to 5.67]
  Serogroup C (Day 360), N=252,240,119,114,133,126 | 11 [8.64 to 13] | 9.02 [7.23 to 11] | 7.53 [5.93 to 9.55] | 4.71 [3.69 to 6.01] | 15 [11 to 21] | 16 [12 to 23]
  Serogroup W (Day 1), N=249,237,119,113,130,124 | 5.5 [4.62 to 6.55] | 5.38 [4.5 to 6.44] | 4.4 [3.52 to 5.51] | 3.43 [2.73 to 4.32] | 6.75 [5.23 to 8.7] | 8.1 [6.25 to 11]
  Serogroup W (Day 360), N=249,237,119,113,130,124 | 42 [35 to 50] | 7.57 [6.33 to 9.07] | 36 [28 to 46] | 4.95 [3.83 to 6.4] | 49 [38 to 62] | 11 [8.75 to 14]
  Serogroup Y (Day 1), N=250,239,118,113,132,126 | 3.29 [2.9 to 3.73] | 3.4 [2.99 to 3.87] | 3.04 [2.62 to 3.53] | 2.56 [2.2 to 2.98] | 3.53 [2.91 to 4.27] | 4.39 [3.61 to 5.35]
  Serogroup Y (Day 360), N=250,239,118,113,132,126 | 27 [22 to 33] | 5.29 [4.34 to 6.45] | 24 [19 to 31] | 3.42 [2.65 to 4.43] | 30 [23 to 40] | 7.82 [5.86 to 10]

9. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Vaccination in Children Aged 2 to 10 Years
Description: Safety and tolerability of a single dose of MenACWY-CRM conjugate vaccine compared to the safety and tolerability of a single dose of licensed MenACWY-PS vaccine when administered to healthy children 2 to 10 years of age.
Time Frame: Day 1 to 7 post vaccination
Population: Analysis was done on safety population i.e. all randomized subjects who received a vaccination and who had follow up safety data.
Measure: Number; unit: Subjects
Groups:
- MenACWY-CRM (2-5 Years Old); MenACWY-CRM (6-10 Years Old): Subjects received one dose of investigational MenACWY-CRM conjugate vaccine
- MenACWY-PS (2-5 Years Old); MenACWY-PS (6-10 Years Old): Subjects received one dose of licensed MenACWY-PS vaccine
Arm/Group | MenACWY-CRM (2-5 Years Old) | MenACWY-PS (2-5 Years Old) | MenACWY-CRM (6-10 Years Old) | MenACWY-PS (6-10 Years Old)
Number analyzed (Participants) | 151 | 153 | 157 | 157
Subjects
  Local reactions | 56 | 37 | 70 | 50
  Injection site pain | 43 | 30 | 57 | 43
  Injection site erythema | 23 | 11 | 26 | 9
  Injection site induration | 17 | 5 | 26 | 6
  Systemic reactions | 55 | 45 | 39 | 28
  Change in eating habits, N=145,150 | 18 | 16 | NA | NA
  Sleepiness | 25 | 24 | NA | NA
  Irritability | 29 | 26 | NA | NA
  Vomiting | 12 | 6 | NA | NA
  Diarrhea | 11 | 6 | NA | NA
  Chills, N=156, 157 | NA | NA | 13 | 5
  Nausea, N=156, 157 | NA | NA | 6 | 6
  Malaise, N=156, 157 | NA | NA | 12 | 9
  Myalgia, N=156, 157 | NA | NA | 12 | 4
  Arthralgia, N=151,153,156,157 | 3 | 7 | 5 | 3
  Headache, N=151,153,156,157 | 6 | 3 | 29 | 17
  Other | 40 | 31 | 37 | 23
  Stayed at home due to reactions, N=146,151,154,156 | 6 | 5 | 6 | 3
  Analg./antipyr. med. used, N=150,152,157,157 | 38 | 28 | 36 | 23

10. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Vaccination in Toddlers Aged 12 to 23 Months
Description: Safety and tolerability of a single dose of MenACWY-CRM conjugate vaccine when administered in healthy toddlers (12-15 months old), alone or concomitantly with PnC and when administered in healthy toddlers (16-23 months old), alone or concomitantly with DTaP.
Time Frame: Day 1 to 7 post vaccination
Population: Analysis was done on safety population.
Measure: Number; unit: Subjects
Groups:
- MenACWY-CRM (12-15 Months); MenACWY-CRM (16-23 Months): Subjects received one dose of investigational MenACWY-CRM conjugate vaccine
- MenACWY-CRM + PnC (12-15 Months): Subjects received one dose of investigational MenACWY-CRM conjugate vaccine concomitantly with PnC
- MenACWY-CRM + DTaP (16-23 Months): Subjects received one dose of investigational MenACWY-CRM conjugate vaccine concomitantly with DTaP
Arm/Group | MenACWY-CRM (12-15 Months) | MenACWY-CRM + PnC (12-15 Months) | MenACWY-CRM (16-23 Months) | MenACWY-CRM + DTaP (16-23 Months)
Number analyzed (Participants) | 74 | 71 | 71 | 73
Subjects
  Local reactions | 37 | 29 | 40 | 35
  Injection site reaction tenderness | 15 | 17 | 19 | 18
  Injection site reaction erythema | 29 | 17 | 30 | 25
  Injection site reaction induration | 16 | 13 | 16 | 10
  Systemic reactions | 47 | 50 | 51 | 50
  Change in eating habits, N=74,70,71,72 | 11 | 20 | 13 | 18
  Sleepiness | 22 | 32 | 21 | 25
  Persistent crying, N=74,70,71,72 | 1 | 3 | 4 | 4
  Irritability | 36 | 40 | 33 | 32
  Vomiting | 1 | 2 | 4 | 5
  Diarrhea | 10 | 11 | 20 | 16
  Other | 35 | 44 | 25 | 41
  Analgesic/antipyretic medicine used | 35 | 44 | 25 | 41

11. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs) After Vaccination in Children Aged 2 to 10 Years
Description: as for outcome 9
Time Frame: Day 1- Day 360 (throughout the study)
Population: Analysis was done on safety population.
Measure: Number; unit: Subjects
Arm/Group | MenACWY-CRM (2-5 Years Old) | MenACWY-PS (2-5 Years Old) | MenACWY-CRM (6-10 Years Old) | MenACWY-PS (6-10 Years Old)
Number analyzed (Participants) | 151 | 153 | 157 | 157
Subjects
  Any AE | 56 | 43 | 45 | 33
  Possibly or probably related AEs | 6 | 7 | 15 | 9
  SAEs | 2 | 1 | 0 | 0
  AEs leading to premature withdrawal | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Vaccination in Toddlers Aged 12 to 23 Months
Description: as for outcome 10
Time Frame: Day 1- Day 360 (Throughout the study)
Population: Analysis was done on safety population.
Measure: Number; unit: Subjects
Groups:
- MenACWY-CRM (12-15 Months Old); MenACWY-CRM (16-23 Months): Subjects received one dose of investigational MenACWY-CRM conjugate vaccine
- MenACWY-CRM + PnC (12-15 Months Old): Subjects received one dose of investigational MenACWY-CRM conjugate vaccine in concomitant with PnC
- MenACWY-CRM + DTaP (16-23 Months): Subjects received one dose of investigational MenACWY-CRM conjugate vaccine in concomitant with DTaP
Arm/Group | MenACWY-CRM (12-15 Months Old) | MenACWY-CRM + PnC (12-15 Months Old) | MenACWY-CRM (16-23 Months) | MenACWY-CRM + DTaP (16-23 Months)
Number analyzed (Participants) | 74 | 71 | 71 | 73
Subjects
  Any AE | 35 | 33 | 25 | 30
  Possibly or probably related AEs | 6 | 1 | 1 | 4
  AEs leading to premature withdrawal | 0 | 0 | 0 | 1
  SAEs | 2 | 3 | 3 | 2

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs), AEs leading to premature withdrawal and any medically significant AEs were collected from Day 1 to 360
Groups:
- MenACWY-PS (6-10 Years Old): Subjects received one dose of the licensed MenACWY-CRM polysaccharide vaccine.
- MenACWY-PnC (12-15 Months Old): Subjects received one dose of the investigational MenACWY-CRM conjugate vaccine administered concomitantly with pneumococcal conjugate vaccine.
- MenACWY+DTaP (16-23 Months Old): Subjects received one dose of the investigational MenACWY-CRM conjugate vaccine administered concomitantly with DTaP vaccine.
- MenACWY-PS (3-5 Years Old): Children aged 3 to 5 years receiving MenACWY-PS from the first part of the study (Menomune not licensed in US in children under 2 years of ages) served as controls for the 12-23-months-old part two toddlers.
Arm/Group | MenACWY (2-5 Years Old) | MenACWY-PS (2-5 Years Old) | MenACWY (6-10 Years Old) | MenACWY-PS (6-10 Years Old) | MenACWY (12-15 Months Old) | MenACWY-PnC (12-15 Months Old) | MenACWY (16-23 Months Old) | MenACWY+DTaP (16-23 Months Old) | MenACWY-PS (3-5 Years Old)
Serious Adverse Events (participants affected / at risk) | 2/151 | 1/153 | 0/157 | 0/157 | 2/74 | 3/71 | 3/71 | 2/73 | 1/100
Other Adverse Events (participants affected / at risk) | 82/151 | 69/153 | 81/157 | 64/157 | 64/74 | 61/71 | 62/71 | 59/73 | 40/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY (2-5 Years Old) (N=151) | MenACWY-PS (2-5 Years Old) (N=153) | MenACWY (6-10 Years Old) (N=157) | MenACWY-PS (6-10 Years Old) (N=157) | MenACWY (12-15 Months Old) (N=74) | MenACWY-PnC (12-15 Months Old) (N=71) | MenACWY (16-23 Months Old) (N=71) | MenACWY+DTaP (16-23 Months Old) (N=73) | MenACWY-PS (3-5 Years Old) (N=100)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APPENDICITIS PERFORATED (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EMPYEMA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PERITONITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FEBRILE CONVULSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY (2-5 Years Old) (N=151) | MenACWY-PS (2-5 Years Old) (N=153) | MenACWY (6-10 Years Old) (N=157) | MenACWY-PS (6-10 Years Old) (N=157) | MenACWY (12-15 Months Old) (N=74) | MenACWY-PnC (12-15 Months Old) (N=71) | MenACWY (16-23 Months Old) (N=71) | MenACWY+DTaP (16-23 Months Old) (N=73) | MenACWY-PS (3-5 Years Old) (N=100)
DIARRHOEA (Gastrointestinal disorders) | 12 | 6 | 0 | 0 | 10 | 12 | 20 | 17 | 4
TEETHING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 7 | 2 | 0 | 3 | 0
VOMITING (Gastrointestinal disorders) | 13 | 6 | 0 | 1 | 1 | 4 | 5 | 6 | 2
CHILLS (General disorders) | 0 | 0 | 13 | 5 | 0 | 0 | 0 | 0 | 0
CRYING (General disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 4 | 0
INJECTION SITE ERYTHEMA (General disorders) | 23 | 11 | 26 | 9 | 29 | 17 | 30 | 25 | 5
INJECTION SITE INDURATION (General disorders) | 17 | 5 | 26 | 6 | 16 | 13 | 16 | 10 | 2
INJECTION SITE PAIN (General disorders) | 43 | 30 | 57 | 43 | 15 | 18 | 19 | 18 | 22
MALAISE (General disorders) | 0 | 0 | 12 | 9 | 0 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 12 | 10 | 3 | 4 | 7 | 4 | 4 | 6 | 7
CROUP INFECTIOUS (Infections and infestations) | 2 | 1 | 0 | 0 | 2 | 5 | 1 | 2 | 0
OTITIS MEDIA (Infections and infestations) | 4 | 3 | 0 | 0 | 8 | 5 | 0 | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 6 | 4 | 4 | 10 | 6 | 0 | 5 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 12 | 4 | 0 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 7 | 3 | 29 | 18 | 0 | 0 | 0 | 0 | 3
SOMNOLENCE (Nervous system disorders) | 25 | 24 | 0 | 0 | 22 | 32 | 21 | 25 | 13
EATING DISORDER (Psychiatric disorders) | 18 | 16 | 0 | 0 | 11 | 20 | 13 | 18 | 9
IRRITABILITY (Psychiatric disorders) | 29 | 26 | 0 | 0 | 36 | 40 | 33 | 32 | 14
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1 | 2 | 4 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days